CLINICAL TRIAL: NCT03323320
Title: Evaluation of Patient's Knowledge of Their NACO Treatment
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: AOD
Record Dates: First submitted 2017-10-24; First posted 2017-10-27 (Actual); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Anticoagulant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
More than one million of patient receive anti vitamine K treatment which is the main cause of hospitalization. About 50 000 patient receive direct oral anticoagulant .

The aim is to evaluate the patient's level of knowledge about their anticoagulant treatment and specially about the side effect

ELIGIBILITY:
Inclusion Criteria:

* patient with AOD treatment
* capable to answer to questionnaire
* with or without antivitamin K

Exclusion Criteria:

* dementia
* cognitive trouble
* refusing participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients under AOD treatment in GHPSJ (hospitalization and consultation)
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2016-12-05 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
questionnaire score >80% | Day 1
  it's a questionnaire about anticoagulant treatment ; each question has a score ans for the study investigators calculate the total

CONTACTS AND LOCATIONS:
Overall Officials: Romain CADOR, MD, Study Director — GHPSJ
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France